CLINICAL TRIAL: NCT04273295
Title: Massage With Senna-based Laxatives Versus Senna-based Laxatives in Managing Overflow Retentive Stool Incontinence in Pediatrics
Brief Title: Massage With Senna-based Laxatives Versus Senna-based Laxatives in Managing Overflow Retentive Stool Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002277
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Massage
Keywords: Constipation; Laxatives; Massage
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: First group receives senna-based laxatives . Second group managed by abdominal massage with senna-based laxatives. Evaluation of outcome of two groups as regard to continence and radiological study.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (No Intervention): This group receives senna-based laxatives.
- the study group (Experimental): This group managed by abdominal massage with senna-based laxatives.
  Interventions: Other: Abdominal massage

INTERVENTIONS:
Other: Abdominal massage — The patients lying in comfortable relaxed supine position and physiotherapist performed slow circular clockwise movements on the abdomen, throw tangential pushing, with digital pulp, slow and gradual pressure, with fingers inclination 45 degree. The pressure applied to the abdomen on each point for 1 min, beginning with the ascending colon, transverse colon, descending colon and sigmoid; this sequence was repeated approximately 15 min. The therapist teaches the parents this technique and asked them to apply at home 3 times / day for 15 min.
  Arms: the study group

SUMMARY:
This study aimed to evaluate the effect of abdominal massage with senna-based laxative in managing overflow retentive stool incontinence in pediatrics.

DETAILED DESCRIPTION:
Much attention has been devoted to children with overflow retentive stool incontinence (ORSI) by the pediatric surgeons, as the referral of such cases from pediatric facilities is constantly increasing. An important initial step in managing these children is the exclusion of Hirschsprung's disease starting by water-soluble contrast enema.

Conservative management of ORIS is generally successful. The aim of the treatment is to achieve and maintain regular bowel movements free of symptoms Laxatives remain the mainstay of maintenance therapy of ORSI; yet, there is no standard laxative therapy despite the varieties of medication currently available. New information to these queries can be beneficial to medical staff involved in managing overflow retentive stool incontinence in pediatrics, Possibly it may add new guideline of treatment with more good result , short time and decrease the laxative dose.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with ORSI according to Rome III criteria
* Contrast enema suggestive of fecal loading
* the absence of anatomic, physiologic or pathologic reason for their constipation

Exclusion Criteria:

* radiological suspicion of Hirschsprung's disease,
* anorectal malformation,
* mechanical obstruction,
* failed to comply with the offered treatment (mainly if cramping abdominal pain or vomiting occurred),
* Required bowel surgery.
* spina bifida, spinal cord injury,

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
starting dose | starting dose was assessed at day 0.
  the effective starting dose at the begining of treatment.
starting dose | starting dose was assessed at day 180.
  the effective starting dose at the begining of treatment.
end dose | end dose was assessed at day 0.
  the effective ending dose (maintenance dose) at the end of treatment.
end dose | end dose was assessed at day 180.
  the effective ending dose (maintenance dose) at the end of treatment.
time till not soiling | time till not soiling was assessed at day 0.
  Stool soiling (encopresis) happens in children who are toilet trained. It's when they accidentally leak feces (poop) into their underwear. Constipation is one of many causes of stool soiling. Other causes include irritable bowel syndrome or when a child is fearful of the bathroom.
time till not soiling | time till not soiling was assessed at day 180.
  Stool soiling (encopresis) happens in children who are toilet trained. It's when they accidentally leak feces (poop) into their underwear. Constipation is one of many causes of stool soiling. Other causes include irritable bowel syndrome or when a child is fearful of the bathroom.

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, Ph.D, Principal Investigator — South Valley University; Nezar A. Abo Halawa, Ph.D, Principal Investigator — South Valley University; Mohammed E. Ali, Ph.D, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levitt MA, Pena A. Minimally invasive treatment of fecal incontinence and constipation in children. Minerva Chir. 2010 Apr;65(2):223-34. PMID 20548277
- [Background] Turnbull GK, Lennard-Jones JE, Bartram CI. Failure of rectal expulsion as a cause of constipation: why fibre and laxatives sometimes fail. Lancet. 1986 Apr 5;1(8484):767-9. doi: 10.1016/s0140-6736(86)91783-6. PMID 2870270
- [Background] Turan N, Ast TA. The Effect of Abdominal Massage on Constipation and Quality of Life. Gastroenterol Nurs. 2016 Jan-Feb;39(1):48-59. doi: 10.1097/SGA.0000000000000202. PMID 26825564
- [Result] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Result] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Result] Voskuijl WP, Heijmans J, Heijmans HS, Taminiau JA, Benninga MA. Use of Rome II criteria in childhood defecation disorders: applicability in clinical and research practice. J Pediatr. 2004 Aug;145(2):213-7. doi: 10.1016/j.jpeds.2004.04.050. PMID 15289770
- [Result] Voskuijl W, de Lorijn F, Verwijs W, Hogeman P, Heijmans J, Makel W, Taminiau J, Benninga M. PEG 3350 (Transipeg) versus lactulose in the treatment of childhood functional constipation: a double blind, randomised, controlled, multicentre trial. Gut. 2004 Nov;53(11):1590-4. doi: 10.1136/gut.2004.043620. PMID 15479678
- [Result] Nurko S, Youssef NN, Sabri M, Langseder A, McGowan J, Cleveland M, Di Lorenzo C. PEG3350 in the treatment of childhood constipation: a multicenter, double-blinded, placebo-controlled trial. J Pediatr. 2008 Aug;153(2):254-61, 261.e1. doi: 10.1016/j.jpeds.2008.01.039. Epub 2008 Mar 19. PMID 18534221
- [Result] Le Blanc-Louvry I, Costaglioli B, Boulon C, Leroi AM, Ducrotte P. Does mechanical massage of the abdominal wall after colectomy reduce postoperative pain and shorten the duration of ileus? Results of a randomized study. J Gastrointest Surg. 2002 Jan-Feb;6(1):43-9. doi: 10.1016/s1091-255x(01)00009-9. PMID 11986017
- [Result] Weerapong P, Hume PA, Kolt GS. The mechanisms of massage and effects on performance, muscle recovery and injury prevention. Sports Med. 2005;35(3):235-56. doi: 10.2165/00007256-200535030-00004. PMID 15730338
- [Result] McClurg D, Lowe-Strong A. Does abdominal massage relieve constipation? Nurs Times. 2011 Mar 29-Apr 4;107(12):20-2. PMID 21520798
- [Result] Liu Z, Sakakibara R, Odaka T, Uchiyama T, Yamamoto T, Ito T, Hattori T. Mechanism of abdominal massage for difficult defecation in a patient with myelopathy (HAM/TSP). J Neurol. 2005 Oct;252(10):1280-2. doi: 10.1007/s00415-005-0825-9. Epub 2005 May 20. No abstract available. PMID 15895308
- [Result] Lamas K, Lindholm L, Stenlund H, Engstrom B, Jacobsson C. Effects of abdominal massage in management of constipation--a randomized controlled trial. Int J Nurs Stud. 2009 Jun;46(6):759-67. doi: 10.1016/j.ijnurstu.2009.01.007. Epub 2009 Feb 12. PMID 19217105

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT04273295/Prot_SAP_000.pdf